CLINICAL TRIAL: NCT06934694
Title: Effect of Instrument-Assisted Soft Tissue Mobilization on Gastrocnemius Muscle Stiffness and Ankle Dorsiflexion Range of Motion
Brief Title: Effect of Instrument-Assisted Soft Tissue Mobilization on Gastrocnemius Stiffness and Ankle Range of Motion
Acronym: IASTM-Gastro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Žiga Kozinc, PhD, Assistant professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IASTM_Gastro
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Muscle Stiffness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM (Experimental): Participants in this arm will receive a single session of instrument-assisted soft tissue mobilization (IASTM) applied to the gastrocnemius muscle. The treatment will be performed using a standardized protocol that includes longitudinal and cross-friction strokes with a stainless-steel tool. The intervention is designed to target the superficial and deep layers of the gastrocnemius and will be delivered for a total of approximately 5 minutes. Post-treatment assessments of muscle stiffness and ankle dorsiflexion range of motion will be conducted immediately following the intervention.
  Interventions: Device: Instrument-Assisted Soft Tissue Mobilization
- Control (No Intervention)

INTERVENTIONS:
Device: Instrument-Assisted Soft Tissue Mobilization — Participants will receive a single session of instrument-assisted soft tissue mobilization (IASTM) applied to the gastrocnemius muscle using a stainless-steel instrument. The treatment consists of longitudinal and transverse strokes targeting both the medial and lateral heads of the muscle. The procedure will be performed by a trained clinician, following a standardized protocol lasting approximately 5 minutes. The goal is to induce mechanical and neuromodulatory effects on muscle tissue. This intervention is designed to assess acute changes in muscle stiffness (via shear-wave elastography) and ankle dorsiflexion range of motion (via the weight-bearing lunge test).
  Arms: IASTM

SUMMARY:
This study will examine whether a technique called instrument-assisted soft tissue mobilization (IASTM) can reduce stiffness in the calf muscle (gastrocnemius) and improve ankle mobility. Muscle stiffness will be measured using a specialized ultrasound method called shear-wave elastography, while ankle range of motion will be assessed using the weight-bearing lunge test. Healthy volunteers will participate in this study, and measurements will be taken before and after a single IASTM treatment. The aim is to determine if this manual therapy technique can produce immediate changes in muscle properties and joint flexibility.

DETAILED DESCRIPTION:
This interventional study aims to evaluate the acute effects of instrument-assisted soft tissue mobilization (IASTM) on the stiffness of the gastrocnemius muscle and ankle dorsiflexion range of motion. Muscle stiffness will be quantified using shear-wave elastography (SWE), a non-invasive ultrasound technique that measures tissue mechanical properties in real time. Ankle dorsiflexion range of motion will be assessed using the weight-bearing lunge test with the knee extended, a reliable functional measure of ankle mobility.

Participants will undergo baseline measurements followed by a standardized IASTM intervention targeting the gastrocnemius muscle. Post-treatment assessments will be conducted immediately afterward to capture acute changes. The study is designed to improve understanding of how IASTM influences muscle mechanical properties and functional joint mobility. Findings may have implications for the clinical use of IASTM in both rehabilitation and performance contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Healthy individuals without current lower limb injury
* No history of surgery to the ankle, knee, or calf
* Able to perform the weight-bearing lunge test without assistance
* Willing to refrain from intense lower-limb exercise 24 hours before testing

Exclusion Criteria:

* Current or recent (past 3 months) lower limb musculoskeletal pain or injury
* Known neuromuscular or vascular disorders affecting the lower extremity
* Use of medications affecting muscle tone or flexibility within 48 hours prior to testing
* Previous adverse reactions to manual therapy or IASTM
* Skin lesions, bruising, or conditions over the gastrocnemius that contraindicate IASTM
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Muscle stiffness | Baseline and Immediately Post-Intervention
  Stiffness of the gastrocnemius muscle will be measured using shear-wave elastography (SWE), a non-invasive ultrasound technique that quantifies the shear modulus of soft tissue. Measurements will be performed with the participant in a prone position, with the ankle in a standardized neutral position, to ensure consistency. The shear modulus (in kilopascals) will be used as the primary metric of muscle stiffness.
  Time Frame:

SECONDARY OUTCOMES:
Ankle Dorsiflexion Range of Motion | Baseline and Immediately Post-Intervention
  Ankle dorsiflexion range of motion will be assessed using the weight-bearing lunge test with the knee extended. The distance from the great toe to the wall will be recorded at the point where the heel remains in contact with the floor while the knee touches the wall. This test is a reliable and functional assessment of gastrocnemius-related ankle flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No